CLINICAL TRIAL: NCT03741647
Title: Prognostic Significance of Sleep Apnea in Non Small Cell Lung Cancer
Brief Title: Sleep Apnea and Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmad Abbas, Principal investigator &lecturer of chest disases zagazig university, Zagazig University
Other Study IDs: ZU-IRB #:4791/30-7-2018
Record Dates: First submitted 2018-09-21; First posted 2018-11-15 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Locally Advanced Non Small Cell Lung Cancer
MeSH Terms: interventions — Polysomnography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: sleep study and blood sample — full night polysomnographic study and blood sample to detect some genetic issues

SUMMARY:
cases of locally advanced non small cell lung cancer (diagnosed by PET/CT scan and histopathological confirmation) will be screened for sleep disorders by Epworth sleepiness scale then confirmed by full night polysomnographic study. Blood sample to detect some genetic determinants will be withdrawn

ELIGIBILITY:
Inclusion Criteria:

* patients with locally advanced non small cell lung cancer

Exclusion Criteria:

* unable or refuse to perform sleep study
* metastatic cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - patients with locally advanced non small cell lung cancer diagnosed, managed and followed up in clinical oncology department, zagazig university hospitals
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
assessment Response to treatment | 6 weeks from ending therapy
  CT chest/pelvi-abdomen with contrast (evaluation using RECIST criteria)
confirmed Response to treatment | 4 weeks from assessment response
  CT chest/pelvi-abdomen with contrast (evaluation using RECIST criteria)

SECONDARY OUTCOMES:
Progression Free Survival | 3 months from confirmed response to treatment
  CT chest/pelvi-abdomen with contrast (evaluation using RECIST criteria)
Progression Free Survival | 6 months from confirmed response to treatment
  CT chest/pelvi-abdomen with contrast (evaluation using RECIST criteria)
Progression Free Survival | 9 months from confirmed response to treatment
  CT chest/pelvi-abdomen with contrast (evaluation using RECIST criteria)
Progression Free Survival | 12 months from confirmed response to treatment
  CT chest/pelvi-abdomen with contrast (evaluation using RECIST criteria)
Overall survival | 3 months after enrollment
  regular patient follow up visit
Overall survival | 6 months after enrollment
  regular patient follow up visit
Overall survival | 9 months after enrollment
  regular patient follow up visit
Overall survival | 12 months after enrollment
  regular patient follow up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad Abbas, Zagazig, Asharqia, Egypt